CLINICAL TRIAL: NCT00511641
Title: Quality of Life Associated With a Low-Risk Screening Program for Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID01-693
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Cancer Screening; Quality of Life; Questionnaire; Screening; Survey
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Risk OVCA: Patient that is participating in an ovarian cancer (OVCA) screening program.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires lasting up to 30 minutes.
  Other Names: Survey

SUMMARY:
The goal of this research study is to learn more about how women feel about an ovarian cancer screening program that involves getting a blood test to measure CA 125 levels. This includes finding out about women's quality of life and whether they are concerned or worried about their risk of developing cancer. This study also seeks to find out whether elevated CA 125 levels affect participants in terms of cancer worries or concerns.

DETAILED DESCRIPTION:
Participants in this study will be asked to complete several questionnaires. Participants will be able to fill out the questionnaires in the clinic or if necessary, they can complete them at home. Pre-addressed and stamped envelopes will be provided to mail back if they are completed at home. The questionnaires involve quality of life issues, concerns or worries about cancer risk and beliefs about cancer. It will take 30 minutes or less to complete the questionnaires.

The completed questionnaires can be returned to the research nurse or if the participant prefers or they can be returned to the researchers in the self-addressed stamped envelope that is provided.

This is an investigational study. This study will involve 2400 women who are participating in an ovarian cancer screening program. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women enrolled on protocol ID01-022

   * Women > 50 years of age
   * Postmenopausal (> 12 months amenorrhea)
   * Willingness to return to clinic for annual blood tests, or earlier if indicated
   * Willingness to undergo transvaginal ultrasound if indicated
2. Women who speak and read English

Exclusion Criteria:

1. Women ineligible to be enrolled on protocol ID01-022

   * Prior removal of both ovaries
   * Active non-ovarian malignancy
   * Women who have a history of non-ovarian malignancy will be eligible if they have no persistent or recurrent disease and have not received treatment for > 12 months. They will not be excluded if they are on tamoxifen.
   * High-risk for ovarian cancer due to familial predisposition as defined by the following:

     * Known mutation in BRCA1 or BRCA2
     * Two first or second degree relatives with either ovarian cancer or pre-menopausal breast cancer
     * Ashkenazi Jewish ethnicity with one first degree or two second degree relatives with pre-menopausal breast or ovarian cancer, or if patient herself has had breast cancer.
2. Women who do not speak or read English

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female UT MDACC Patients, over 50 years of age, participating in an ovarian cancer screening program.
Sampling Method: Non-Probability Sample
Enrollment: 1342 (Actual)
Dates: Start 2002-02-12 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Mean Scores on Each Quality of Life Instrument (Surveys) | Baseline quality of life data collected, and if/when return to clinic due to abnormal test results.
  Descriptive, written, self-report, quality of life instruments used.

SECONDARY OUTCOMES:
To find out whether elevated CA 125 levels affect participants in terms of cancer worries or concerns. | 8 Years

CONTACTS AND LOCATIONS:
Overall Officials: Diane C. Bodurka, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org